CLINICAL TRIAL: NCT05547477
Title: Continuous EMG Measurements in Children With Asthma During Sleep
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, Job van der Palen, Research Coordinator, Medisch Spectrum Twente
Other Study IDs: R22.068
Record Dates: First submitted 2022-09-09; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Asthma in Children; Electromyography; Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to investigate whether electromyography of the diaphragm during sleep in asthmatic children can be used to objectively monitor asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Paediatrician diagnosed asthma or bronchial hyperresponsiveness
* Aged 4 till 18
* Admitted to the paediatric ward of Medisch Spectrum Twente

Exclusion Criteria:

* Admittance to the ICU
* Patient has ICD or pacemaker
* Parents and/or patient cannot understand or speak Dutch
* Does not fit in one of the available Hexoskin shirts

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators aim to include 20 paediatric patients with paediatrician diagnosed asthma of bronchial hyperresponsiveness, admitted to the paediatric ward of Medisch Spectrum Twente.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Breathing registration in sleep using electromyography | From admittance to the ward, up to 12 hours
  Amplitude of the EMG signal will be used to obtain breathing waveforms.

SECONDARY OUTCOMES:
Prediction of asthma exacerbations | After inclusion of all subjects, up to 3 months
  A machine learning model will be applied to be able to predict an asthma exacerbation before it occurs